CLINICAL TRIAL: NCT03651856
Title: A Pilot Study of Atomoxetine for Freezing of Gait in Parkinson's Disease
Brief Title: Atomoxetine for Freezing of Gait in Parkinson's Disease
Acronym: ATMFOG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014009
Record Dates: First submitted 2018-07-02; First posted 2018-08-29 (Actual); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Parkinson's Disease; Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atomoxetine (Experimental): Atomoxetine 40mg daily for 2 weeks uptitration Atomoxetine 40mg BID for 4 weeks Atomoxetine 40mg daily for 1 week weaning off
  Interventions: Drug: ATM FOG in PD

INTERVENTIONS:
Drug: ATM FOG in PD — open label pilot study on atomoxetine 40mg BID on patients with Parkinson's disease and Freezing of Gait

SUMMARY:
Subjects are being asked to participate in this study to determine the safety and effectiveness of a drug called atomoxetine in the treatment of freezing of gait for Parkinson's Disease patients. Atomoxetine (ATM) is an approved drug currently on the market for the treatment of attention deficit. It works to increase the amount of norepinephrine (a chemical in the brain that helps keep us awake and alert) in our brain. ATM has not been approved by the Food and Drug Administration (FDA) to be used in the treatment of PD, but has been found to be well tolerated in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Idiopathic Parkinson's Disease according to UK Brain Bank Criteria, Hoehn and Yahr stage 2-4
2. A positive response to item 14 of the UPDRS, part 2.
3. Age range 18-80
4. Ability to walk a minimum of 20 feet without assistive device and with one observed freezing episode which may be triggered by visual cue
5. Letter of medical clearance by primary care physician dated within preceding 2 months of subject's initial active study visit.
6. Stable on PD medications for ≥ 3 months

   -

Exclusion Criteria:

1. Intolerance to drug class
2. Mini-Mental Status Examination <26/30
3. No observable episodes of freezing of gait despite common visual cues
4. Not on stable PD medications for 3 months
5. Subjects who whose gait disturbance is due to other conditions not related to PD or FOG.
6. Current use of monoamine oxidase inhibitor (MAO-I)
7. Hypersensitivity to drug class
8. Narrow angle glaucoma
9. Pheochromocytoma
10. Severe cardiovascular disorders, i.e. patients with pre-existing conditions that would be expected to deteriorate if their heart rate or blood pressure were to increase in a clinically significant manner (e.g. 15-20 mmHg increase in blood pressure or 20 beats per minute in heart rate).
11. Patients with uncontrolled hypertension.
12. Patients with a history of symptomatic tachyarrhythmias.
13. Presence of uncontrolled depression and suicidal ideation.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo J Revuelta, DO, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: Count of Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Evaluate the safety of Atomoxetine 40mg bid in PD patients with FOG (Freezing of Gait)
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 10
Participants
  Increase in Creatine | 3
  Worsening Fog (Freezing of Gait) | 1
  Diarrhea | 1
  Worsening Dyskinesia | 1
  Nausea | 1
  Mild Jitters | 1

ADVERSE EVENTS:
Arm/Group | Atomoxetine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=10)
Increase in Creatine (Blood and lymphatic system disorders) | 3 (3)
Worsening Fog (Freezing of Gait) (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Worsening Dyskinesia (Nervous system disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Mild Jitters (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes